CLINICAL TRIAL: NCT06336746
Title: Effects of Steep Trendelenburg and Pneumoperitoneum on Cardiac Performance During Robotic-assisted Surgery in Patients With Normal and Low Ejection Fraction.
Brief Title: Cardiac Performance During Steep Trendelenburg Position in Patients Undergoing Robotic Surgery Surgery.
Status: Recruiting | Type: Observational
Sponsor: Karlstad Central Hospital (Other)
Responsible Party: Principal Investigator, Ragnar Henningsson, Associate Professor, Karlstad Central Hospital
Other Study IDs: RHenningsson
Record Dates: First submitted 2023-12-12; First posted 2024-03-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure, Systolic; Robotic Surgery
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with Preoperative EF: 50% or higher: Patients included will be examined with Transthoracic Echocardiography preoperatively and Ejection Fraction (EF) measured.
  Interventions: Device: Esophageal Doppler
- Patients with Preoperative EF: 45% or lower: Patients included will be examined with Transthoracic Echocardiography preoperatively and Ejection Fraction (EF) measured.
  Interventions: Device: Esophageal Doppler
- Patients without intrathecal bupivacain and morphine.: The routine is that all patient receive an intrathecal injection of morphine and bupivacain before start of anesthesia. Patients who have contraindications for spinal anesthesia will be collected in this group.
  Interventions: Device: Esophageal Doppler

INTERVENTIONS:
Device: Esophageal Doppler — Esophageal Doppler: measuring cardiac performance. INVOS: measuring regional saturation of the brain.
  Other Names: InVivo Optical Spectroscopy INVOS

SUMMARY:
The field of robotic-assisted laparoscopic surgery increases all the time. Older and more fragile patients which are not suitable for major open surgery could be scheduled for robotic- assisted surgery. The peroperative anesthesiological challenges and stresses during this type of surgery could anyway be even more prominent.

The extreme positioning of patients during robotic surgery in the pelvis, often 30 degrees head down tilting (Trendelenburg positioning), should increase the work load of the heart significantly. There are no studies concerning fragile patients with heart failure during these conditions.

In this study the circulatory effects in patients with normal heart function and preexisting heart failure will be studied during robotic surgery in extreme Trendelenburg positioning

During surgery the work load and performance of the heart will be monitored using an esophageal doppler and optical spectrophotometry measuring regional saturation of the brain. This study can identify patients at risk of developing critical circulatory failure during this type of surgery.

DETAILED DESCRIPTION:
BACKGROUND:

The development of robotic-assisted laparoscopic surgery is rapid. It is at least more gentle than open surgery to the patient. During certain types of robotic-surgery i.e. prostatectomies and hysterectomies deep down in the small pelvis the surgeons need to tilt the patient in a steep Trendelenburg (30 degrees head down) position and insufflate CO2 (carbon dioxide) gas into the stomach to reach and visualize the organs properly.

According to the law of gravity this entails that the blood inside the vessels is pressed backwards against the pumping heart and afterload increases. To be able to withhold the flow of blood to our vital organs the performance of our heart is challenged. Besides carbon dioxide is blown into the stomach, which even more increases the workload of the heart. There is a substantial risk of acute heart failure during these manoeuvres especially in patients with preexisting heart failure.

There are very few studies investigating these problems. Earlier studies have only investigated the effects in healthy ASA (American Society of Anesthesiologists) 1-2 patients.

AIM:

This study will investigate how patients with known systolic heart failure manage this strain which is included in this new developing type of robotic surgery compared to patients with normal heart function.

METHOD:

1. Included patients undergo an echocardiographic investigation before surgery and will be classified in 2 groups: a) Normal systolic function b) Decreased systolic function defined as Ejection Fraction (EF) 45% or lower.
2. After start of anesthesia all patients receive an esophageal doppler and the output values of cardiac stroke volume (SV); cardiac Index (CI), systemic vascular resistance (SVR); pulse pressure variation(PPV), stroke Volume variation (SVV) Peak Velocity (PV)and Flow Time Corrected (FTc) are recorded as well as standard routine parameters during anesthesia. With INVOS (In Vivo Optical Spectroscopy) regional oxygen saturation of the front lobes of the brain is measured.
3. This procedure is repeated after start of Trendelenburg position 30 degrees head down, at the start of pneumoperitoneum and at the return to supine position.
4. The effects of robotic assisted surgery between patients with normal EF compared to patients with EF 45% or lower will be compared.

THE IMPORTANCE OF THIS STUDY:

The increasing field of robotic-assisted surgery, which often results in shorter and less complicated postoperative care will enable older and more fragile patients to be available for surgery. In contrast these patients encounter new cardiovascular challenges during the anesthesia and extreme positioning surgery.

It is therefore most important to be aware of these physiological challenges and how to handle them. This study will also show which patients are not suitable for robotic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive Patients Scheduled for Robotic Surgery with Trendelenburg positioning.

-

Exclusion Criteria:

1. Age <18;
2. Dementia,
3. Not able to give written consent -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive Patients scheduled for robotic surgery in Tendelenburg positioning.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Stroke Volume during Trendelenburg position and pneumoperitoneum. | During 15 minutes after reaching position.
  Esophageal Doppler Monitoring

SECONDARY OUTCOMES:
% Change of Systemic Vascular Resistance;PulsePressureVariation; Peak Velocity; Stroke Volume Variation and FlowTimeCorrected | During 15 minutes after reaching position
  Esophageal Doppler Monitoring
% change in regional brain saturation rSO2 during Trendelenburg position and pneumooperitoneum. | During 15 min after reaching position.
  INVivoOpticalSpectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Dpt of Anesthesiology&Intensive Care; Central Hospital of Karlstad, Karlstad, Värmland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided